CLINICAL TRIAL: NCT02227706
Title: A Prospective, Randomized, Controlled Study Evaluating EVICEL® Fibrin Sealant as an Adjunct to Haemostasis During Abdominal, Retroperitoneal, Pelvic or Thoracic (Non-Cardiac) Surgery in Paediatric Patients
Brief Title: The Paediatric EVICEL® Soft Tissue and Parenchymal Organ Bleeding Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ethicon, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 400-12-006; 2013-003401-26 (EudraCT Number)
Record Dates: First submitted 2014-08-26; First posted 2014-08-28 (Estimated); Results first posted 2020-08-31 (Actual); Last update posted 2020-08-31 (Actual); Status verified 2020-08

CONDITIONS: Hemorrhage; Soft Tissue Bleeding
Keywords: Fibrin Sealant; Hemostatics; Coagulants
MeSH Terms: conditions — Hemorrhage | interventions — Fibrin Tissue Adhesive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- EVICEL® Fibrin Sealant (Experimental): EVICEL® is a human plasma-derived fibrin sealant. EVICEL® consists of two components: a concentrate of Human Clottable Protein (referred to as Biological Component 2; BAC2) and a solution of Human Thrombin. No material of animal origin is present in the product
  Interventions: Biological: EVICEL® Fibrin Sealant
- SURGICEL® Absorbable Hemostat (Active Comparator): SURGICEL® Absorbable Hemostat (oxidized regenerated cellulose) is a sterile absorbable knitted fabric prepared by the controlled oxidation of regenerated cellulose.
  Interventions: Device: SURGICEL® Absorbable Hemostat

INTERVENTIONS:
Biological: EVICEL® Fibrin Sealant — EVICEL® is a human plasma-derived fibrin sealant. EVICEL® consists of two components: a concentrate of Human Clottable Protein (referred to as Biological Component 2; BAC2) and a solution of Human Thrombin. No material of animal origin is present in the product
  Other Names: EVICEL, fibrin sealant
  Arms: EVICEL® Fibrin Sealant
Device: SURGICEL® Absorbable Hemostat — SURGICEL® Absorbable Hemostat (oxidized regenerated cellulose) is a sterile absorbable knitted fabric prepared by the controlled oxidation of regenerated cellulose.
  Other Names: oxidized regenerated cellulose
  Arms: SURGICEL® Absorbable Hemostat

SUMMARY:
To evaluate the safety and effectiveness of EVICEL® Fibrin Sealant (Human) as an adjunct to achieve haemostasis during surgery in paediatric patients.

DETAILED DESCRIPTION:
This is a prospective, randomized, controlled, clinical study comparing EVICEL® to SURGICEL®, as an adjunct to haemostasis when conventional methods of controlling bleeding are ineffective or impractical during surgery in paediatric patients.

At least 40 qualified paediatric subjects with an appropriate mild or moderate Target Bleeding Site (TBS) will be randomized in a 1:1 allocation ratio to either EVICEL® or SURGICEL®. Haemostasis will be assessed at 4, 7 and 10 minutes from randomization.

Enrolment will be staggered by age (as required by the European Medicines Agency (EMA) Paediatric Committee). The first group enrolled will include at least 36 subjects aged ≥1 years to <18 years of age. When enrolment of the first group is complete; enrolment of a subsequent group will commence and include at least 4 subjects from birth (including neonates ≤37 weeks gestation) to <1 years of age.

Subjects will be followed post-operatively through hospital discharge and at 30 days (±14 days) post-surgery.

ELIGIBILITY:
Inclusion Criteria:

* Paediatric subjects birth to <18 years of age, requiring non-emergent laparoscopic or open (through peritoneum or pleura) abdominal, retroperitoneal, pelvic or thoracic (non-cardiac) surgical procedures. i) The first 36 subjects to be enrolled will be subjects ≥1 years to <18 years of age. ii) The next 4 subjects to be enrolled will be subjects birth to <1years of age.
* The subject and/or subject's parent or legal guardian must be willing to give permission for the subject to participate in the trial, and provide written informed consent for the subject. If possible, assent must be obtained from paediatric subjects who possess the intellectual and emotional ability to comprehend the concepts involved in the trial. If the paediatric subject is not able to provide assent (due to age, maturity and/or inability to intellectually and/or emotionally comprehend the trial), the parent/legal guardian's written informed consent for the subject will be acceptable for the subject to be included in the study; and
* Presence of an appropriate mild or moderate bleeding soft tissue or parenchymal organ Target Bleeding Site identified intra-operatively by the surgeon;

Exclusion Criteria:

* Subjects with known intolerance to blood products or to one of the components of the study product or is unwilling to receive blood products;
* Female subjects, who are of childbearing age (i.e. adolescent), who are pregnant or nursing;
* Subject is currently participating or, during the study is planned to participate in any other investigational device or drug trial without prior approval from the Sponsor;
* Subjects who are known, current alcohol and/or drug abusers;
* Subjects admitted for trauma surgery;
* Subjects with any pre or intra-operative findings identified by the surgeon that may preclude conduct of the study procedure;
* Subjects with Target Bleeding Site in an actively infected field (Class III Contaminated or Class IV Dirty or Infected)
* Anastomotic bleeding sites will not be considered for randomization.

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2014-08-01 (Actual); Primary Completion 2019-04-17 (Actual); Study Completion 2019-05-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Kocharian, MD, PhD, Study Director — Ethicon, Inc.
Locations (13):
- Clinical Investigation Site #31, Brussels, Belgium
- Canada (3):
  - Clinical Investigation Site #42, Hamilton, Ontario
  - Clinical Investigation Site #40, Toronto, Ontario
  - Clinical Investigation Site #41, Montreal, Quebec
- United Kingdom (9):
  - Clinical Investigation Site #21, Birmingham
  - Clinical Investigation Site #22, Leeds
  - Clinical Investigation Site #20, Liverpool
  - Clinical Investigation Site #27, London
  - Clinical Investigation Site #23, London
  - Clinical Investigation Site #26, London
  - Clinical Investigation Site #30, Newcastle
  - Clinical Investigation Site #25, Nottingham
  - Clinical Investigation Site #24, Southampton

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were screened up to 21 days prior to surgery and attended a baseline visit within 24 hours of surgery. Both visits took place at a clinic within the hospital where surgery also took place. Subjects were followed until discharge and requested to attend a visit at 30 days (+/- 14 days) post surgery either at the hospital or via telephone.
Pre-assignment Details: Subjects required to meet pre-defined inclusion/exclusion criteria prior to randomization. Subjects required to have an appropriate mild or moderate target bleeding site identified intra-operatively.
  Subjects were excluded if the target bleeding site was in an actively infected field or if the bleeding was at an anastomotic bleeding site.
Groups:
- EVICEL®: EVICEL® is a human plasma derived fibrin sealant consisting of two components: (1) Biologically Active Component 2 (BAC2), a concentrate of human clottable protein (containing mainly human fibrinogen and fribrinectin), and (2) human thrombin.
- SURGICEL®: SURGICEL® Absorbable hemostat is a sterile absorbable knitted fabric prepared by controlled oxidation of regenerated cellulose.
Period: Overall Study
Arm/Group | EVICEL® | SURGICEL®
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | EVICEL® | SURGICEL® | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Full Range); unit: Years] | 9.4 [0.9 to 17.0] | 9.0 [1.0 to 17.0] | 9.2 [0.9 to 17.0]
Age, Customized [Number; unit: Participants]
  Neonate (Birth to 30 Days) | 0 | 0 | 0
  Infants and toddlers (31 days-<24 months) | 5 | 2 | 7
  Children (2-11 years) | 4 | 9 | 13
  Adolescents (12-17 years) | 11 | 9 | 20
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 7 | 18
  Male | 9 | 13 | 22
Race/Ethnicity, Customized [Number; unit: Participants]
  White/Caucasian | 16 | 16 | 32
  Asian | 2 | 2 | 4
  Other | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Absolute Time to Haemostasis
Description: Absolute time to haemostasis, defined as absolute time when there was no detectable bleeding at the Target Bleeding Site (TBS).
Time Frame: From randomisation (identification of appropriate target bleeding site) to final fascial closure (median study procedure time 164.0 minutes [range 47.0 - 506.0 minutes])
Population: Full Analysis Set (all randomized subjects)
Measure: Median (95% Confidence Interval); unit: Minutes
Arm/Group | EVICEL® | SURGICEL®
Number analyzed (Participants) | 20 | 20
Minutes | 4.0 [3.3 to 4.7] | 4.0 [2.9 to 8.1]

2. Secondary Outcome: Number of Participants Achieving Haemostasis at 4 Minutes
Description: Number of participants achieving haemostasis at target bleeding site at 4 minutes. This endpoint is assessing haemostasis at 4 minutes only and not maintenance of haemostasis following this timepoint. As rebleeding may occur between timepoints, subsequent rebleeding (if any) is detailed in treatment failure analysis.
Time Frame: Intra-operatively from randomisation to 4 minutes after randomisation
Population: Full Analysis Set (all randomized subjects)
Measure: Count of Participants; unit: Participants
Arm/Group | EVICEL® | SURGICEL®
Number analyzed (Participants) | 20 | 20
Participants | 16 | 13

3. Secondary Outcome: Number of Participants Achieving Haemostasis at 7 Minutes
Description: Number of Participants Achieving Haemostasis at Target Bleeding Site at 7 Minutes. This endpoint is assessing haemostasis at 7 minutes only and is not affected by haemostasis assessment prior to 7 minutes or maintenance of haemostasis following this 7 minute assessment. As rebleeding may occur between timepoints, subsequent rebleeding (if any) is detailed in treatment failure analysis.
Time Frame: Intra-operatively from randomisation to 7 minutes after randomisation
Population: Full Analysis Set (all randomized subjects)
Measure: Count of Participants; unit: Participants
Arm/Group | EVICEL® | SURGICEL®
Number analyzed (Participants) | 20 | 20
Participants | 20 | 16

4. Secondary Outcome: Number of Participants Achieving Haemostasis at 10 Minutes
Description: Number of Participants Achieving Haemostasis at Target Bleeding Site at 10 Minutes. This endpoint is assessing haemostasis at 10 minutes only and is not affected by haemostasis assessments prior to 10 minutes or maintenance of haemostasis following this 10 minute assessment. As rebleeding may occur between timepoints, subsequent rebleeding (if any) is detailed in treatment failure analysis).
Time Frame: Intra-operatively from randomisation to 10 minutes after randomisation
Population: Full Analysis Set (all randomized subjects)
Measure: Count of Participants; unit: Participants
Arm/Group | EVICEL® | SURGICEL®
Number analyzed (Participants) | 20 | 20
Participants | 19 | 18

5. Secondary Outcome: Incidence of Treatment Failures (Number of Participants)
Description: Defined as haemostasis not achieved within 10 minutes or bleeding requiring treatment other than re-application of the assigned haemostatic adjunct within 10 minutes.
Time Frame: 10 minutes
Population: Full Analysis Set (all randomized subjects) Note: Two subjects in the control arm were haemostatic at the TBS at 10 minutes however they subsequently rebled requiring additional treatment and were conservatively considered a failure for the secondary endpoint of Incidence of Treatment Failures.
Measure: Count of Participants; unit: Participants
Arm/Group | EVICEL® | SURGICEL®
Number analyzed (Participants) | 20 | 20
Participants | 1 | 5

6. Secondary Outcome: Estimated Blood Loss
Description: Blood loss during surgical procedure (includes but not limited to the target bleeding site)
Time Frame: During surgical procedure (first incision to final fascial closure (median study procedure time 164.0 minutes [range 47.0 - 506.0 minutes])
Population: Full Analysis Set (all randomized subjects)
Measure: Median (Full Range); unit: mL
Arm/Group | EVICEL® | SURGICEL®
Number analyzed (Participants) | 20 | 20
mL | 50.0 [0.0 to 2000.0] | 50.0 [0.0 to 400.0]

7. Secondary Outcome: Blood Transfusion
Description: Participants requiring a blood transfusion
Time Frame: From surgical procedure to 30 day (+/-14 day) follow-up visit
Population: Full Analysis Set (all randomized subjects)
Measure: Count of Participants; unit: Participants
Arm/Group | EVICEL® | SURGICEL®
Number analyzed (Participants) | 20 | 20
Participants
  Yes (Blood Transfusion Received) | 7 | 3
  No (Blood Transfusion Not Received) | 13 | 17

8. Secondary Outcome: Participants Receiving a Blood Transfusion
Description: Details of blood products received (if any)
Time Frame: From surgery to 30 day (+/-14 day) follow-up visit
Population: Full Analysis Set (all randomized subjects with data)
Measure: Count of Participants; unit: Participants
Arm/Group | EVICEL® | SURGICEL®
Number analyzed (Participants) | 20 | 20
Participants
  Packed Red Blood Cells 0 Units: number analyzed (Participants) | 7 | 3
  Packed Red Blood Cells 0 Units | 3 | 0
  Packed Red Blood Cells 1 Unit: number analyzed (Participants) | 7 | 3
  Packed Red Blood Cells 1 Unit | 4 | 1
  Packed Red Blood Cells 2 Units: number analyzed (Participants) | 7 | 3
  Packed Red Blood Cells 2 Units | 0 | 2
  Whole Blood 0 Units: number analyzed (Participants) | 7 | 3
  Whole Blood 0 Units | 4 | 3
  Whole Blood 1 Unit: number analyzed (Participants) | 7 | 3
  Whole Blood 1 Unit | 0 | 0
  Whole Blood 2 Units: number analyzed (Participants) | 7 | 3
  Whole Blood 2 Units | 3 | 0
  Fresh Frozen Plasma 0 Units: number analyzed (Participants) | 7 | 3
  Fresh Frozen Plasma 0 Units | 6 | 3
  Fresh Frozen Plasma 1 Unit: number analyzed (Participants) | 7 | 3
  Fresh Frozen Plasma 1 Unit | 0 | 0
  Fresh Frozen Plasma 2 Units: number analyzed (Participants) | 7 | 3
  Fresh Frozen Plasma 2 Units | 1 | 0
  Platelets 0 Units: number analyzed (Participants) | 7 | 3
  Platelets 0 Units | 6 | 3
  Platelets 1 Unit: number analyzed (Participants) | 7 | 3
  Platelets 1 Unit | 1 | 0
  Cryoprecipitates 0 Units: number analyzed (Participants) | 7 | 3
  Cryoprecipitates 0 Units | 7 | 3
  Other 0 Units: number analyzed (Participants) | 7 | 3
  Other 0 Units | 7 | 3

9. Secondary Outcome: Changes in Laboratory Parameters Haemoglobin and Mean Corpuscular Haemoglobin Concentration
Description: Laboratory parameter changes from baseline to post operative hospital discharge (Haemoglobin and Mean Corpuscular Haemoglobin Concentration)
Time Frame: Baseline (within 21 days prior to surgery) to Hospital Discharge (within 72 hours of discharge)
Population: Safety Set (all subjects who received treatment)
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | EVICEL® | SURGICEL®
Number analyzed (Participants) | 20 | 20
g/L
  Haemoglobin g/L: number analyzed (Participants) | 20 | 18
  Haemoglobin g/L | -13.2 (21.5) | -10.6 (8.9)
  Mean Corpuscular Haemoglobin Concentration g/L: number analyzed (Participants) | 16 | 17
  Mean Corpuscular Haemoglobin Concentration g/L | -5.3 (6.7) | -3.4 (11.9)

10. Secondary Outcome: Changes in Laboratory Parameters Haematocrit
Description: Change in red blood cell proportion in volume in the blood from baseline to post operative hospital discharge
Time Frame: Baseline (within 21 days prior to surgery) to Hospital Discharge (within 72 hours of discharge)
Population: Safety Set (all subjects who received treatment)
Measure: Mean (Standard Deviation); unit: L/L
Arm/Group | EVICEL® | SURGICEL®
Number analyzed (Participants) | 20 | 20
L/L | -0.0 (0.0) | -0.0 (0.0)

11. Secondary Outcome: Changes in Laboratory Parameters Platelet Count and White Cell Count
Description: Laboratory parameter changes from baseline to post operative hospital discharge
Time Frame: Baseline (within 21 days prior to surgery) to Hospital Discharge (within 72 hours)
Population: Safety Set (all subjects who received treatment)
Measure: Mean (Standard Deviation); unit: Cells*10^9/L
Arm/Group | EVICEL® | SURGICEL®
Number analyzed (Participants) | 20 | 20
Cells*10^9/L
  Platelet Count *10^9/L: number analyzed (Participants) | 20 | 18
  Platelet Count *10^9/L | 27.4 (159.3) | 7.6 (96.3)
  White Blood Cell Count *10^9/L: number analyzed (Participants) | 20 | 18
  White Blood Cell Count *10^9/L | 2.0 (5.2) | 1.4 (4.3)

12. Secondary Outcome: Changes in Laboratory Parameters Red Blood Cell Count
Description: Laboratory parameter changes from baseline to post operative hospital discharge
Time Frame: Baseline (within 21 days prior to surgery) to Hospital Discharge (within 72 hours of discharge)
Population: Safety Set (all subjects who received treatment)
Measure: Mean (Standard Deviation); unit: Cells*10^12/L
Arm/Group | EVICEL® | SURGICEL®
Number analyzed (Participants) | 20 | 20
Cells*10^12/L | -0.3 (0.5) | -0.4 (0.4)

13. Secondary Outcome: Changes in Laboratory Parameters Mean Corpuscular Haemoglobin
Description: Laboratory parameter changes from baseline to post operative hospital discharge
Time Frame: Baseline (within 21 days prior to surgery) to Hospital Discharge (within 72 hours of discharge)
Population: Safety Set (all subjects who received treatment)
Measure: Mean (Standard Deviation); unit: pg
Arm/Group | EVICEL® | SURGICEL®
Number analyzed (Participants) | 20 | 20
pg | -0.1 (1.1) | 0.2 (0.9)

14. Secondary Outcome: Changes in Laboratory Parameters Mean Corpuscular Volume
Description: Laboratory parameter changes from baseline to post operative hospital discharge
Time Frame: Baseline (within 21 days prior to surgery) to Hospital Discharge (within 72 hours of discharge)
Population: Safety Set (all subjects who received treatment)
Measure: Mean (Standard Deviation); unit: f/L
Arm/Group | EVICEL® | SURGICEL®
Number analyzed (Participants) | 20 | 20
f/L | 0.9 (2.6) | 1.5 (3.2)

15. Secondary Outcome: Changes in Laboratory Parameters Neutrophils, Lymphocytes, Monocytes, Eosinophils and Basophils
Description: Laboratory parameter changes in volume from baseline to post operative hospital discharge (Neutrophils, Lymphocytes, Monocytes, Eosinophils and Basophils)
Time Frame: Baseline (within 21 days prior to surgery) to Hospital Discharge (within 72 hours of discharge)
Population: Safety Set (all subjects who received treatment)
Measure: Mean (Standard Deviation); unit: Percent Volume
Arm/Group | EVICEL® | SURGICEL®
Number analyzed (Participants) | 20 | 20
Percent Volume
  Neutrophils %: number analyzed (Participants) | 20 | 18
  Neutrophils % | 9.0 (17.1) | 10.1 (19.4)
  Lymphocytes %: number analyzed (Participants) | 20 | 18
  Lymphocytes % | -7.2 (13.1) | -11.6 (17.3)
  Monocytes %: number analyzed (Participants) | 20 | 18
  Monocytes % | -0.8 (6.4) | 1.5 (2.1)
  Basophils %: number analyzed (Participants) | 20 | 18
  Basophils % | -0.1 (0.4) | -0.3 (0.4)

16. Secondary Outcome: Changes in Laboratory Parameters Activated Partial Thromboplastin Time and Prothrombin Time
Description: Laboratory parameter changes from baseline to post operative hospital discharge (Activated Partial Thromboplastin Time and Prothrombin Time)
Time Frame: Baseline (within 21 days prior to surgery) to Hospital Discharge (within 72 hours of discharge)
Population: Safety Set (all subjects who received treatment)
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | EVICEL® | SURGICEL®
Number analyzed (Participants) | 20 | 20
Seconds
  Activated Partial Thromboplastin Time seconds: number analyzed (Participants) | 13 | 10
  Activated Partial Thromboplastin Time seconds | -0.9 (4.2) | -2.2 (4.2)
  Prothrombin Time seconds: number analyzed (Participants) | 13 | 12
  Prothrombin Time seconds | 0.7 (3.0) | 0.1 (1.3)

17. Secondary Outcome: Changes in Laboratory Parameters International Normalised Ratio
Description: Standardized measurement of the change in blood clotting time from baseline to post operative hospital discharge
Time Frame: Baseline (within 21 days prior to surgery) to Hospital Discharge (within 72 hours of discharge)
Population: Safety Set (all subjects who received treatment)
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | EVICEL® | SURGICEL®
Number analyzed (Participants) | 20 | 20
Ratio | 0.1 (0.2) | -0.0 (0.1)

18. Other Pre Specified Outcome: Number of Participants With a Thrombotic Event
Description: Number of Participants with a Thrombotic Event.
Time Frame: From randomisation up to 30 days (+/- 14 days) following surgery
Population: Safety Set (all subjects who received treatment)
Measure: Count of Participants; unit: Participants
Arm/Group | EVICEL® | SURGICEL®
Number analyzed (Participants) | 20 | 20
Participants
  Number of subjects with thrombotic events | 0 | 0

19. Other Pre Specified Outcome: Number of Participants With an Adverse Event Related to Re-bleeding at Target Bleeding Site
Description: Number of Participants with an Adverse Event Related to Re-bleeding at Target Bleeding Site.
Time Frame: From randomisation to 30 days (+/- 14 days) following surgery
Population: Safety Set (all subjects who received treatment)
Measure: Count of Participants; unit: Participants
Arm/Group | EVICEL® | SURGICEL®
Number analyzed (Participants) | 20 | 20
Participants
  Subjects with AE related to re-bleeding at TBS | 1 | 2

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from point of randomisation, during the procedure, throughout hospital admission and until completion of the 30 day (+/-14 day) follow up visit.
Description: Additional adverse event collection information:
  Since post operative pain is an expected outcome of this type of surgery, for purposes of this study, only exacerbations of expected post operative pain based on the Investigator's judgment were reported as an AE.
Arm/Group | EVICEL® | SURGICEL®
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 4/20 | 3/20
Other Adverse Events (participants affected / at risk) | 18/20 | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EVICEL® (N=20) | SURGICEL® (N=20)
Varicella (Infections and infestations) | 1 (1) | 0 (0) — Chicken Pox
Brain Injury (Nervous system disorders) | 1 (1) | 0 (0) — Hypoxic Brain Injury
Clostridium difficile infection (Infections and infestations) | 1 (1) | 0 (0)
Ureteral stent removal (Surgical and medical procedures) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Castleman's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EVICEL® (N=20) | SURGICEL® (N=20)
Coagulopathy (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 2 (2)
Tachycardia (Cardiac disorders) | 3 (3) | 6 (6)
Conjunctivitis (Eye disorders) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 5 (5) | 3 (3)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 4 (4)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mucous stools (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 2 (2)
Teething (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 6 (6)
Chest pain (General disorders) | 0 (0) | 1 (1)
Device occlusion (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 8 (9) | 6 (7)
Swelling (General disorders) | 0 (0) | 1 (1)
Candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Orchitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Post procedural infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Viral infection (Infections and infestations) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 7 (8) | 5 (5)
Wound complication (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Wound secretion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood potassium decreased (Investigations) | 0 (0) | 1 (1)
C-reactive protein increased (Investigations) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 1 (1) | 2 (2)
Oxygen saturation decreased (Investigations) | 1 (1) | 2 (3)
Respiratory rate decreased (Investigations) | 1 (1) | 0 (0)
Respiratory rate increased (Investigations) | 1 (1) | 0 (0)
Urine output decreased (Investigations) | 2 (2) | 0 (0)
White blood cell count increased (Investigations) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemic syndrome (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Polydipsia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Convulsion (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 2 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1)
Polyuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Testicular pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Neonatal aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Livedo reticularis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Wound drainage (Surgical and medical procedures) | 0 (0) | 1 (1)
Haemorrhage (Vascular disorders) | 1 (1) | 2 (2)
Hypertension (Vascular disorders) | 1 (1) | 2 (2)
Hypotension (Vascular disorders) | 2 (2) | 2 (3)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication based on the results obtained at the trial site (or group of sites) shall not be made before the first multi-centre publication.

During the review period of a proposed publication, the Sponsor is entitled to request that publication be delayed for a period of up to six months from the date of first submission to the Sponsor to enable the Sponsor to take steps to protect its proprietary information and/or Intellectual Property Rights and Know How.

DOCUMENTS (2):
  • Study Protocol (2018-01-08): https://cdn.clinicaltrials.gov/large-docs/06/NCT02227706/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-01): https://cdn.clinicaltrials.gov/large-docs/06/NCT02227706/SAP_001.pdf